CLINICAL TRIAL: NCT00101829
Title: An Open-Label, One Arm, Phase I Safety Study of Anti-CD20 Antibody (Rituximab, Rituxan) Therapy in the Treatment of Primary Sjogren's Syndrome
Brief Title: Anti-CD20 Antibody Therapy for Sjogren's Syndrome
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Autoimmunity Centers of Excellence (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DAIT ASJ01
Record Dates: First submitted 2005-01-13; First posted 2005-01-14 (Estimated); Last update posted 2017-10-20 (Actual); Status verified 2017-10

CONDITIONS: Sjogren's Syndrome
Keywords: Autoimmune Diseases
MeSH Terms: conditions — Sjogren's Syndrome; Autoimmune Diseases | interventions — Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Rituximab Treatment (Experimental): Participants will receive rituximab at study entry and at Week 2
  Interventions: Drug: Rituximab

INTERVENTIONS:
Drug: Rituximab — 1000 mg intravenous infusion
  Other Names: Rituxan

SUMMARY:
The purpose of this study is to determine the safety of the anti-CD20 antibody rituximab in treating patients with Sjogren's syndrome (SS). Rituximab is a laboratory-made antibody currently used to treat some kinds of lymphoma. Rituximab may also help people with SS, a disease of the immune system. However, the safety of rituximab in SS patients must first be established.

DETAILED DESCRIPTION:
SS is the second most common autoimmune disease; it is caused by immune cells attacking and destroying the glands that produce tears and saliva, and occurs more often in women than in men. Currently, there are no established disease-modifying treatments for SS. Traditional treatment strategies for SS primarily address dryness symptoms. Rituximab targets the CD20 antigen on the surface of B cells, and was approved in 1997 for the treatment of patients with low-grade or follicular B-cell non-Hodgkin's lymphoma. In a small study, rituximab was also shown to relieve the symptoms of rheumatoid arthritis. Because SS is associated with the development of B cell-related cancers and rituximab has the potential to treat autoimmune disease, rituximab may alleviate the symptoms of SS. This study will evaluate the safety of rituximab in people with SS.

This study will last 1 year. At 4 and 2 weeks before the start of the study, patients will undergo medical and medication history assessment, a physical exam, blood and urine collection, rheumatologic evaluation, an eye exam, and salivary gland tests. The screening visit 4 weeks before study start will also include an electrocardiogram (ECG), a chest x-ray, and a tuberculosis exam. Patients will receive IV rituximab at study entry and at Week 2; blood collection will occur prior to infusion and post-infusion for pharmacokinetics studies. There will be 6 follow-up study visits that will occur at Weeks 4, 8, 14, 26, 30, and 52. Blood and urine collection; a physical exam; rheumatologic evaluation; and eye, skin, and salivary gland tests will occur at selected study visits.

ELIGIBILITY:
Inclusion Criteria:

* Weighs at least 40 kg (88.2 lbs)
* Meets European criteria proposed by the American-European Consensus Group for primary Sjogren's syndrome
* Has 1 or more of the following symptoms of Sjogren's syndrome: fatigue; joint pain; peripheral neuropathy; interstitial lung disease; leukocytoclastic vasculitis; renal tubular acidosis; interstitial nephritis; severe parotid swelling; or other extraglandular manifestations causing organ system dysfunction
* Agrees to use acceptable methods of contraception during the study and for 12 months after the end of treatment

Exclusion Criteria:

* Active infection
* Chronic or persistent infection which might be worsened by immunosuppressive treatment (e.g., HIV, hepatitis B or C, tuberculosis [TB])
* Known coronary artery disease, significant cardiac arrhythmias, or severe congestive heart failure (New York Heart Association class III or IV)
* Current use of anticoagulants
* Prior use of rituximab
* Cyclophosphamide treatment within 24 weeks prior to screening
* Certain medications that may cause dry mouth
* Cytotoxic therapy with azathioprine, cyclosporine, methotrexate, or mycophenolate mofetil within 4 weeks prior to screening
* Etanercept within 4 weeks prior to screening
* Adalumimab within 8 weeks prior to screening
* Infliximab within 12 weeks prior to screening
* Prednisone at greater than 10 mg/day within 2 weeks prior to screening. Patients who have their steroid doses tapered to 10 mg/day or less within 2 weeks of screening are not excluded.
* Definitive diagnosis of another autoimmune rheumatologic disease (e.g., systemic lupus erythematosus, scleroderma, rheumatoid arthritis)
* History of alcohol or substance abuse
* History of immunoglobulin E (IgE)-mediated or non-IgE-mediated hypersensitivity
* Known anaphylaxis to mouse-derived proteins
* History of head and neck radiation therapy
* History of sarcoidosis (inflammation of unknown cause occurring in the lymph nodes, lungs, liver, eyes, skin, or other tissues)
* History of graft-versus-host disease
* History of cancer. Patients who have had resected basal or major squamous cell carcinoma, cervical dysplasia, or in situ cervical cancer Grade I within the last 5 years prior to study entry are not excluded.
* History of positive PPD without documentation of treatment for TB infection or chemoprophylaxis for TB exposure
* Live vaccines within the 3 months prior to study entry
* Severe pulmonary disease. Patients who do not have undue fatigue or dyspnea following ordinary physical activity are not excluded.
* Psychiatric disorder precluding informed consent
* Inability or unwillingness to follow study requirements
* Any current condition or treatment that, in the opinion of the investigator, may interfere with the study
* Pregnancy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2004-04; Primary Completion 2006-08 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
Count of Participants with Rituximab Related Grade 3 or higher AEs | Throughout study
  The study site will grade the severity of adverse events (AEs) experienced by the study participants according to the criteria set forth in the National Cancer Institute's Common Toxicity Criteria for Adverse Events Version 3.0 (published June 10, 2003).

CONTACTS AND LOCATIONS:
Overall Officials: Philip L. Cohen, MD, Principal Investigator — Rheumatology Division, University of Pennsylvania; E. William St. Clair, MD, Principal Investigator — Division of Rheumatology and Immunology, Duke University Medical Center
Locations (2):
- United States (2):
  - Duke University Medical Center, Durham, North Carolina
  - University of Pennsylvania, Philadelphia, Pennsylvania

REFERENCES:
- [Background] Boye J, Elter T, Engert A. An overview of the current clinical use of the anti-CD20 monoclonal antibody rituximab. Ann Oncol. 2003 Apr;14(4):520-35. doi: 10.1093/annonc/mdg175. PMID 12649096
- [Background] Cheson BD. Rituximab: clinical development and future directions. Expert Opin Biol Ther. 2002 Jan;2(1):97-110. doi: 10.1517/14712598.2.1.97. PMID 11772344
- [Background] Looney RJ, Anolik J, Sanz I. B cells as therapeutic targets for rheumatic diseases. Curr Opin Rheumatol. 2004 May;16(3):180-5. doi: 10.1097/00002281-200405000-00003. PMID 15103242
- [Result] St Clair EW, Levesque MC, Prak ET, Vivino FB, Alappatt CJ, Spychala ME, Wedgwood J, McNamara J, Moser Sivils KL, Fisher L, Cohen P; Autoimmunity Centers of Excellence. Rituximab therapy for primary Sjogren's syndrome: an open-label clinical trial and mechanistic analysis. Arthritis Rheum. 2013 Apr;65(4):1097-106. doi: 10.1002/art.37850. PMID 23334994
- See also: National Institute of Allergy and Infectious Diseases (NIAID) — https://www.niaid.nih.gov
- Available data/document: Individual Participant Data Set: SDY961 — http://www.immport.org/immport-open/public/study/study/displayStudyDetail/SDY961 — ImmPort study identifier is SDY961
- Available data/document: Study Protocol: SDY961 — http://www.immport.org/immport-open/public/study/study/displayStudyDetail/SDY961 — ImmPort study identifier is SDY961
- Available data/document: Study summary, -design, -adverse event(s), - assessments, -medications, -demographics, -files , -laboratory tests, et al.: SDY961 — http://www.immport.org/immport-open/public/study/study/displayStudyDetail/SDY961 — ImmPort study identifier is SDY961